CLINICAL TRIAL: NCT04050384
Title: Effect of a Vibratory Stimulus on the Mitigation of Nociception-specific Behavioral and Electroencephalographic Responses to Skin Puncture in Neonates: a Randomized Control Trial
Brief Title: Effect of a Vibratory Stimulus on Mitigating Nociception-specific Responses to Skin Puncture in Neonates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lance M Relland, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Lance M Relland, MD, PhD, Assistant Professor, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB18-00779
Record Dates: First submitted 2018-11-19; First posted 2019-08-08 (Actual); Results first posted 2023-11-29 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Infant, Newborn; Infant, Premature; Pain Perception; Pain Measurement; Pain Management; Electroencephalography
MeSH Terms: conditions — Premature Birth; Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Personnel who code the video recording for behavioral measures and analysis of the electroencephalographic readings will be done in a blinded and/or independent fashion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- No vibratory stimulus before or during heel lance (No Intervention): Baseline measurements and readings after vibration alone will be done, but no vibratory stimulus will be provided immediately preceding or during heel lance.
- Vibratory stimulus before and during heel lance (Experimental): Baseline measurements and readings after vibration alone will be done, as well as a vibratory stimulus that will be provided immediately preceding and during heel lance.
  Interventions: Device: Baby GentleStick

INTERVENTIONS:
Device: Baby GentleStick — The Baby GentleStick is a handheld device that fits and provides vibration to an Owen Mumford Unistik3 Dual lancet. The gentle vibration occurs at 178 Hertz with a free-hanging 0.24 mm range of motion. The device may provide vibration alone and also allow for simultaneous vibration and deployment of the lancet.
  Arms: Vibratory stimulus before and during heel lance

SUMMARY:
The assessment and treatment of pain in neonates remains a challenge. In an effort to improve the quality of care while limiting opioid-related adverse effects, this study aims to determine the efficacy of a non-pharmacological intervention on the mitigation of nociception-specific responses to a skin breaking procedure in term and preterm neonates. Such responses will be measured using behavioral measures as well as with electroencephalography-based methods.

DETAILED DESCRIPTION:
Eligible neonates who are 36-56 weeks post-menstrual age and who are scheduled to undergo a clinically required heel lance will be studied after obtaining appropriate verbal and written consent from the respective parents. Subjects will be monitored during a baseline resting state, during vibratory stimuli alone, and during a heel lance that is randomized to be preceded or not preceded by the vibratory stimulus. The sessions will include time-locked video recordings and electroencephalography using a specialized net of 128 electrodes (Electrical Geodesics Inc., EGI; Eugene, OR). Behavioral and cortical responses will be then be analyzed in a blinded fashion to determine the efficacy of the vibratory intervention, as well as to validate what behavioral responses are most correlated with nociception-specific cortical activity.

ELIGIBILITY:
Inclusion Criteria:

* Neonatal Intensive Care Unit patient
* Between 36 to 56 weeks post-menstrual age
* Medically stable
* Due to have a clinically required bedside heel stick as part of their routine care

Exclusion Criteria:

* Congenital anomalies or abnormalities affecting the brain
* Patient is over 4 months corrected age
* Infants who receive analgesics or sedatives within 72 hours prior to assessment
* Administration of maternal analgesics or sedatives to which the infant may be exposed

Ages: 36 Weeks to 56 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 134 (Actual)
Dates: Start 2018-11-13 (Actual); Primary Completion 2020-01-23 (Actual); Study Completion 2020-01-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lance Relland, MD, PhD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grunau RE, Oberlander T, Holsti L, Whitfield MF. Bedside application of the Neonatal Facial Coding System in pain assessment of premature neonates. Pain. 1998 Jun;76(3):277-286. doi: 10.1016/S0304-3959(98)00046-3. PMID 9718246
- [Background] Maitre NL, Stark AR, McCoy Menser CC, Chorna OD, France DJ, Key AF, Wilkens K, Moore-Clingenpeel M, Wilkes DM, Bruehl S. Cry presence and amplitude do not reflect cortical processing of painful stimuli in newborns with distinct responses to touch or cold. Arch Dis Child Fetal Neonatal Ed. 2017 Sep;102(5):F428-F433. doi: 10.1136/archdischild-2016-312279. Epub 2017 May 12. PMID 28500064
- [Background] Relland LM, Gehred A, Maitre NL. Behavioral and Physiological Signs for Pain Assessment in Preterm and Term Neonates During a Nociception-Specific Response: A Systematic Review. Pediatr Neurol. 2019 Jan;90:13-23. doi: 10.1016/j.pediatrneurol.2018.10.001. Epub 2018 Oct 10. PMID 30449602
- [Derived] Relland LM, Kjeldsen CP, Jeanvoine A, Emery L, Adderley K, Srinivas R, McLoughlin M, Maitre NL. Vibration-based mitigation of noxious-evoked responses to skin puncture in neonates and infants: a randomised controlled trial. Arch Dis Child Fetal Neonatal Ed. 2024 Oct 18;109(6):622-627. doi: 10.1136/archdischild-2023-326588. PMID 38479794

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | No Vibratory Stimulus Before or During Heel Lance | Vibratory Stimulus Before and During Heel Lance
Started | 67 | 67
Completed | 67 | 67
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Total number of final analysis patients may be lower due to attrition of data.
Groups:
- Total: Total of all reporting groups
Arm/Group | No Vibratory Stimulus Before or During Heel Lance | Vibratory Stimulus Before and During Heel Lance | Total
Number analyzed (Participants) | 67 | 67 | 134
Age, Continuous [Median (Inter-Quartile Range); unit: weeks] — Post-conceptional Population: Data attrition is due to background noise in EEG signal.
  weeks
    number analyzed (Participants) | 40 | 41 | 81
    (all) | 39.5 [38.1 to 40.6] | 39.1 [37.6 to 40.6] | 39.4 [37.9 to 40.6]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Analysis was limited to those with a usable EEG signal.
  Participants
    number analyzed (Participants) | 40 | 41 | 81
    Female | 17 | 14 | 31
    Male | 23 | 27 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Analysis was limited to those with a usable EEG signal.
  Participants
    number analyzed (Participants) | 40 | 41 | 81
    Hispanic or Latino | 0 | 1 | 1
    Not Hispanic or Latino | 40 | 40 | 80
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Analysis was limited to those with a usable EEG signal.
  Participants
    number analyzed (Participants) | 40 | 41 | 81
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 2 | 2 | 4
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 3 | 3 | 6
    White | 29 | 31 | 60
    More than one race | 6 | 5 | 11
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — Population: Analysis was limited to those with a usable EEG signal.
  participants
    United States: number analyzed (Participants) | 40 | 41 | 81
    United States | 40 | 41 | 81
Facial Score [Median (Inter-Quartile Range); unit: units on a scale] — The Facial Score in this study is an adaptation of the established Neonatal Facial Coding System (NFCS) such that seven predetermined components of NFCS are assessed to generate a score that could range from 0 to 7 and for which lower to higher values represent better to worse outcomes, respectively. Of note, a zero value score is meaningful and valid in this case, which makes it possible to yield a median value of zero.
  units on a scale | 0 [0 to 1] | 0 [0 to 1] | 0 [0 to 1]

OUTCOME MEASURES:

1. Primary Outcome: Change in Nociception-specific Brain Activity
Description: Electroencephalography (EEG)-based measurements will be done to detect changes in nociception-specific cortical activity. Recordings will be done using a high-density array of 128 electrodes embedded in soft sponges (Electrical Geodesics, Inc. (EGI); Eugene, Oregon, USA) soaked in warm saline and applied to the infant's head to record event-related potentials (ERPs) with a sampling rate of 1000 Hz, filters set to 0.1-400 Hz. As per published protocols, the midline Cz electrode will be used as the reference. Previous studies have also determined the EEG-based nociception-specific response to occur 350-700 ms after the stimulus. Changes in the amplitude of the signal during this time frame is the primary outcome measure.
Time Frame: EEG-based responses are very brief, so the relevant assessment window is 350-700 ms after stimulus
Population: Subjects who had usable, artifact-free EEG data.
Measure: Mean (Standard Deviation); unit: microvolts*milliseconds
Arm/Group | No Vibratory Stimulus Before or During Heel Lance | Vibratory Stimulus Before and During Heel Lance
Number analyzed (Participants) | 40 | 41
microvolts*milliseconds
  Frontal | 17.9 (39.5) | 9.9 (17.1)
  Central | 11.5 (12.1) | 10.2 (6.8)
  Central Parietal | 12.2 (15.4) | 12.0 (12.4)
Statistical Analysis 1: Comparison: No Vibratory Stimulus Before or During Heel Lance vs Vibratory Stimulus Before and During Heel Lance; Test type: Other; p < 0.001, ANCOVA; These analyses apply to the Frontal, Central, and Central-Parietal regions

2. Secondary Outcome: Change in Facial Expression
Description: Components from the Neonatal Facial Coding System (NFCS) use facial actions to monitor pain in newborn infants. Facial actions that occur each score 1 point, while those that do not occur each score 0 points (better outcome). This study applied 7 facial actions and may therefore score between 0 and 7. A higher score (worse outcome) is interpreted as a higher pain intensity. Comparison of median scores between groups will determine the effect of the intervention, which should result in a lower score to represent mitigation of pain.
Time Frame: Assessment of facial expression is done based on video clips that are synchronized with the ERP window of 350-700ms after stimulus
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | No Vibratory Stimulus Before or During Heel Lance | Vibratory Stimulus Before and During Heel Lance
Number analyzed (Participants) | 40 | 41
units on a scale | 4 [2.75 to 5] | 4 [3 to 5]
Statistical Analysis 1: Comparison: No Vibratory Stimulus Before or During Heel Lance vs Vibratory Stimulus Before and During Heel Lance; Test type: Other; p = 0.38, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: From the time of the clinically required lab draw session to the time the lab results were obtained, all occurred within the same day.
Description: This study involved only placing a soft sponge cap on the head +/- applying a vibratory stimulus to the surface of the skin while performing a standard heel stick for clinically required lab draws.
Arm/Group | No Vibratory Stimulus Before or During Heel Lance | Vibratory Stimulus Before and During Heel Lance
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/67
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/67
Other Adverse Events (participants affected / at risk) | 0/67 | 0/67

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-12-19): https://cdn.clinicaltrials.gov/large-docs/84/NCT04050384/Prot_SAP_002.pdf
  • Informed Consent Form (2018-12-19): https://cdn.clinicaltrials.gov/large-docs/84/NCT04050384/ICF_001.pdf